CLINICAL TRIAL: NCT05306353
Title: Combining a CD40L-Binding Protein (VIB4920) With a TNF-alpha Inhibitor for the Treatment of Inadequately Controlled Rheumatoid Arthritis (ITN092AI)
Brief Title: CD40L Antagonism in Rheumatoid Arthritis (RA)
Acronym: CONTROL-RA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is being closed early due to insufficient participant enrollment across study sites.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN092AI
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; VIB4920; TNFi
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VIB4920 Placebo with TNFi (Placebo Comparator): Participants will receive VIB4920 placebo in a blinded fashion intravenously at weeks 0, 2, 4, 8, and 12 and continue all background disease-modifying RA therapy, including the TNFi, through the study period VIB4920 placebo consists of 0.9% normal saline in 250mL bags.
  Interventions: Drug: Placebo for VIB4920
- VIB4920 with TNFi (Experimental): Participants will receive VIB4920 in a blinded fashion intravenously at a dose of 1500 mg at weeks 0, 2, 4, 8, and 12 and continue all background disease-modifying RA therapy, including the TNFi, through the study period
  Interventions: Drug: VIB4920 with TNFi
- VIB4920 without TNFi (Experimental): Participants will stop TNFi after randomization to this arm, and receive VIB4920 in an evaluator-blinded fashion intravenously at a dose of 1500 mg at weeks 0, 2, 4, 8, and 12 while maintaining all other background disease-modifying RA therapy (e.g., methotrexate, hydroxychloroquine, etc.) through the study period. This arm is evaluator blinded (not aware of treatment status), with the participant aware of treatment status but evaluator is not, due to not using a TNFi placebo for this study
  Interventions: Drug: VIB4920 without TNFi

INTERVENTIONS:
Drug: Placebo for VIB4920 — 26 participants will receive VIB4920 placebo administered intravenously at weeks 0, 2, 4, 8, and 12 while continuing background rheumatoid arthritis (RA) therapy including tumor necrosis factor alpha inhibitor (TNFi) (double-blinded)
  Arms: VIB4920 Placebo with TNFi
Drug: VIB4920 with TNFi — 52 participants will receive 1500 mg administered intravenously at weeks 0, 2, 4, 8, and 12 while continuing background rheumatoid arthritis (RA) therapy including Tumor necrosis factor alpha inhibitor (TNFi) (double blinded)
  Arms: VIB4920 with TNFi
Drug: VIB4920 without TNFi — Participants will receive 1500 mg administered intravenously at weeks 0, 2, 4, 8, and 12 but discontinue necrosis factor alpha inhibitor (TNFi) while continuing all other background rheumatoid arthritis (RA) therapy (evaluator-blinded)
  Arms: VIB4920 without TNFi

SUMMARY:
The primary objective is to determine if the addition of a 12-week course of treatment with VIB4920 to TNFi treatment will result in improved clinical disease control in patients with RA who have had an inadequate response to a TNFi.

DETAILED DESCRIPTION:
This study is a phase 2, multi-site, prospective, randomized, placebo-controlled, three-arm [two arms double-blinded, one arm evaluator-blinded (participant is aware of his/her treatment status, but evaluator is not)] trial of VIB4920 in 104 adults with seropositive Rheumatoid arthritis (RA) in the United States. Individuals will be eligible if they have moderate or high disease activity (Simplified Disease Activity Index [SDAI] ≥ 17) despite treatment with a TNFi for at least 12 weeks. All FDA-approved TNFi (including biosimilars) administered subcutaneously utilizing FDA-approved dosing regimens are permitted.

ELIGIBILITY:
Inclusion Criteria:

1. Participant or legally authorized representative must be able to understand and provide informed consent
2. Adults ≥ 18 years of age
3. Diagnosed with RA by fulfilling the ACR/EULAR 2010 Classification Criteria for RA ≥ 6 months prior to screening (Appendix 9)
4. Documented positive test for rheumatoid factor (RF) and/or anti-cyclic citrullinated peptide antibody (ACPA)
5. SDAI ≥ 17
6. At least 4 tender and 4 swollen joints by a 44 joint count (Appendix 5)
7. Receiving treatment with an FDA-approved TNFi (including biosimilars) that is dosed subcutaneously at an FDA-approved dosing regimen for at least 12 weeks.
8. Willing to continue or discontinue treatment with their current TNFi at the same dose depending upon study arm assignment
9. If treated with leflunomide, sulfasalazine, or hydroxychloroquine, must be taking a stable dose for at least 12 weeks
10. If treated with methotrexate, must be taking a stable dose for at least 12 weeks. The following exceptions are permitted within the 12 weeks prior to screening:

    1. Holding methotrexate after COVID-19 vaccination as per American College of Rheumatology guidance (https://rheumatology.org/)
    2. Holding methotrexate for 1 or 2 weeks after influenza vaccination
11. All participants who engage in sexual activity that could lead to pregnancy must agree to use abstinence or an FDA-approved contraception for the duration of the study to prevent pregnancy

Exclusion Criteria:

1. Inability or unwillingness to give written informed consent or comply with the study protocol
2. Prior or ongoing systemic inflammatory or autoimmune disease (other than RA and secondary Sjögren's syndrome) requiring or potentially requiring other systemic immunomodulatory therapy during the 40-week study period
3. Use of glucocorticoid and/or disease-modifying therapies as specified below:

   1. Prior treatment with any B cell depleting therapy (e.g., rituximab)
   2. Treatment with other biologic therapy (i.e., not targeting TNF-α), including abatacept, tocilizumab, or sarilumab within the previous 12 weeks
   3. Treatment with a JAK inhibitor within the previous 12 weeks
   4. Concurrent use of methotrexate and leflunomide in combination
   5. Prednisone > 10 mg a day or equivalent glucocorticoid use within the previous 4 weeks
   6. Intramuscular, intra-articular, or intravenous glucocorticoids within the previous 4 weeks
   7. Other immunomodulatory medications within the previous 12 weeks except for methotrexate, leflunomide, sulfasalazine, or hydroxychloroquine
4. Lack of any subjective or objective clinical response (i.e., complete non-responder) to treatment with the current TNFi, in the opinion of the study investigator based on available documentation in the medical record and/or history provided by the patient and/or referring rheumatologist
5. Use of an investigational agent including VIB4920 in the past 30 days or 5 half-lives, whichever is longer
6. History of a severe allergy, hypersensitivity reaction, or infusion reaction to any component of the VIB4920 formulation
7. History of Felty's syndrome
8. History of interstitial lung disease with FVC < 70% predicted, DLCO < 70% predicted, or requiring supplemental oxygen
9. Arterial or deep venous thromboembolism including pulmonary embolism in the prior two years
10. Infection:

    a. Evidence of current or prior infection with hepatitis B, as indicated by a positive test for the hepatitis B surface antigen (HBsAg) or a positive test for the hepatitis B core antibody (HBcAb) b. Positive HCV serology unless treated with an anti-viral regimen resulting in a sustained virologic response (undetectable viral load 24 weeks after cessation of therapy) c. Evidence of HIV infection d. Evidence of active tuberculosis, untreated or incompletely treated latent tuberculosis, or recent close contact with a person who has active tuberculosis e. Positive QuantiFERON-TB Gold, QuantiFERON-TB Gold Plus, or T-SPOT-TB test without history of previous treatment for active or latent TB f. Indeterminate QuantiFERON-TB Gold, QuantiFERON-TB Gold Plus, or T-SPOT.TB test which remains indeterminate on repeat testing, and any of the following additional required screening which indicates an increased risk of TB infection: i. History of tuberculosis exposure ii. History of travel to an area where tuberculosis is endemic iii. Findings on chest radiograph suggestive of prior exposure to tuberculosis (e.g., granulomas or apical scarring) obtained at screening or within the past 3 months iv. Positive purified protein derivative (PPD) skin test for tuberculosis obtained in the past 3 months, either obtained at screening or within the past 3 months v. Prior history of a positive QuantiFERON-TB Gold, QuantiFERON-TB Gold Plus, T- SPOT.TB, or purified protein derivative (PPD) test without history of previous treatment for latent TB g. Symptoms of presumed or documented SARS-CoV-2 infection in the past 30 days h. More than one episode of herpes zoster in the past 12 months

    i. An opportunistic infection in the past 12 months j. Acute or chronic infection, including current use of suppressive systemic anti-microbial therapy for chronic or recurrent bacterial or fungal infection, hospitalization for treatment of infection in the past 60 days, or parenteral anti-microbial (including anti-bacterial, anti-viral, or anti-fungal agents) use in the past 60 days for infection k. History of bronchiectasis with recurrent pulmonary infections
11. History of a primary immunodeficiency disorder
12. Vaccination with a live vaccine within the past 30 days
13. Women who are pregnant or breast-feeding
14. White Blood Cell (WBC) count < 3.0 x 103/μl
15. Absolute neutrophil count < 1.5 x 103/μl
16. Hemoglobin < 9 g/dL
17. Platelet count < 100 x 103/μl
18. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2x the upper limit of normal (ULN)
19. History of malignant neoplasm within the last 5 years, except for basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the uterine cervix treated locally
20. Current, diagnosed mental illness or current, diagnosed or self-reported drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements
21. Any new or uncontrolled condition occurring within the past 12 weeks which, in the judgment of the investigator, could interfere with participation in the trial (e.g., diabetes mellitus with HbA1c ≥ 9.0%, myocardial infarction, or stroke)
22. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study
23. Inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving low disease activity by Simplified Disease Activity Index (SDAI) | Week 16
  Defined by a Simplified Disease Activity Index (SDAI) <= 11
  Participants who escalate their disease-modifying therapy or take any prohibited medications for treatment of RA prior to Week 16 are considered to have failed the primary endpoint. The primary analysis will compare the primary endpoint between the two blinded study arms: VIB4920 with TNFi and VIB4920 placebo with TNFi study arms

SECONDARY OUTCOMES:
Proportion of participants who achieve sustained remission | Week 16 to Week 40
  Defined by Simplified Disease Activity Index (SDAI) <= 3.3
Proportion of participants achieving low disease activity by Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) | Week 16
  Defined by Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) <= 3.2
Proportion of participants achieving remission defined by SDAI | Week 16
  Defined by Simplified Disease Activity Index (SDAI) <= 3.3. Participants who escalate their disease-modifying therapy or take prohibited medications for treatment of their RA prior to week 16 are considered to have failed this secondary endpoint
Proportion of participants achieving remission defined by DAS28-CRP | Week 16
  Defined by Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) < 2.6. Participants who escalate their disease-modifying therapy or take prohibited medications for treatment of their Rheumatoid Arthritis (RA) prior to week 16 are considered to have failed this secondary endpoint
The proportion of participants achieving an ACR20 response | Week 16
The proportion of participants achieving an ACR50 response | Week 16
The proportion of participants achieving an ACR70 response | Week 16
The proportion of participants achieving an ACR20 response | Week 40
The proportion of participants achieving an ACR50 response | Week 40
The proportion of participants achieving an ACR 70 response | Week 40
Time to first occurrence of low disease activity as defined by SDAI | Week 0 to Week 40
  Defined by SDAI <= 11; for participants who fail to achieve low disease activity or remission prior to escalating their disease-modifying therapy or taking a prohibited medication for treatment of RA, we will assume low disease activity and remission is not achievable.
Time to first occurrence of low disease activity as defined by DAS28-CRP | Week 0 to Week 40
  Defined by Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) <= 3.2; for participants who fail to achieve low disease activity or remission prior to escalating their disease-modifying therapy or taking a prohibited medication for treatment of RA, we will assume low disease activity and remission is not achievable.
Time to first occurrence of remission as defined by SDAI | Week 0 to Week 40
  Defined by Simplified Disease Activity Index (SDAI) <= 3.3; for participants who fail to achieve low disease activity or remission prior to escalating their disease-modifying therapy or taking a prohibited medication for treatment of RA, we will assume low disease activity and remission is not achievable.
Time to first occurrence of remission as defined by DAS28-CRP | Week 0 to Week 40
  Defined by Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) < 2.6; for participants who fail to achieve low disease activity or remission prior to escalating their disease-modifying therapy or taking a prohibited medication for treatment of RA, we will assume low disease activity and remission is not achievable.
Time to loss of low disease activity defined by SDAI | Week 16
  Defined by Simplified Disease Activity Index (SDAI) > 11 for the subset of individuals achieving low disease activity by the SDAI criteria. Participants who escalate their disease-modifying therapy or take prohibited medications for treatment of their RA will be considered to have lost the low disease activity or remission response
Time to loss of low disease activity defined by DAS28-CRP | Week 16
  Defined by Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) > 3.2 for the subset of individuals achieving low disease activity by the DAS28-CRP criteria. Participants who escalate their disease-modifying therapy or take prohibited medications for treatment of their RA will be considered to have lost the low disease activity or remission response
Time to loss of remission defined by SDAI | Week 16
  Defined by Simplified Disease Activity Index (SDAI) > 3.3 for the subset of individuals achieving remission by the SDAI criteria. Participants who escalate their disease-modifying therapy or take prohibited medications for treatment of their RA will be considered to have lost the low disease activity or remission response
Time to loss of remission defined by DAS28-CRP | Week 16
  Defined by DAS28-CRP >= 2.6 for the subset of individuals achieving remission by the DAS28-CRP criteria. Participants who escalate their disease-modifying therapy or take prohibited medications for treatment of their RA will be considered to have lost the low disease activity or remission response
Longitudinal trends in Simplified Disease Activity Index (SDAI) | Week 0 to Week 40
Longitudinal trends in Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) | Week 0 to Week 40
Change in the Health Assessment Questionnaire - Disability Index (HAQ-DI) | Week 0 to 16
Change in the Health Assessment Questionnaire - Disability Index (HAQ-DI) | Week 0 to 40
Change in Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) Profile scores | Week 0 to Week 40
Change in Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) Profile scores | Week 0 to 16
Incidence of grade 2 or higher adverse events (AEs) | Week 0 to Week 40
  Liver chemistry abnormalities will be graded using protocol specific criteria, defined relative to the upper limit of normal (ULN):
  * Aspartate aminotransferase [AST] increased: Grade 2: > 3.0x ULN - 5.0x ULN, Grade 3: > 5.0x ULN - 20.0x ULN, Grade 4: > 20.0x ULN
  * Alanine aminotransferase [ALT] increased: Grade 2: > 3.0x ULN - 5.0x ULN, Grade 3: > 5.0x ULN - 20.0x ULN, Grade 4: > 20.0x ULN
  * Alkaline phosphatase [ALP] increased: Grade 2: > 2.5x ULN - 5.0x ULN, Grade 3: > 5.0x ULN - 20.0x ULN, Grade 4: > 20.0x ULN
  * Blood bilirubin increased: Grade 2: > 1.5x ULN - 3.0x ULN, Grade 3: > 3.0x ULN - 10.0x ULN, Grade 4: > 10.0x ULN
  All other AEs will be graded according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence of serious adverse events | Week 0 to Week 40
  An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or Sponsor (DAIT/NIAID), it results in any of the following outcomes (21 CFR 312.32(a)):
  1. Death.
  2. A life-threatening event: An AE or SAR is considered "life-threatening" if, in the view of either the investigator or Sponsor (DAIT/NIAID), its occurrence places the participant at immediate risk of death. It does not include an AE or SAR that, had it occurred in a more severe form, might have caused death.
  3. Inpatient hospitalization or prolongation of existing hospitalization.
  4. Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
  5. Congenital anomaly or birth defect.
Incidence of adverse events of special interest (AESI) | Week 0 to Week 40
  The following are considered Adverse Events of Special Interest (AESI):
  * Anaphylaxis and grade 3 or higher hypersensitivity reactions
  * Grade 3 or higher infusion reactions
  * AST or ALT >3xULN with serum total bilirubin > 2xULN (Hy's Law)
  * Grade 3 or higher infection
  * Opportunistic infections including but not limited to reactivation of latent viral infections, invasive fungal infections, and TB
  * Malignant neoplasm
  * Immune complex disease

CONTACTS AND LOCATIONS:
Overall Officials: Eugene William St. Clair, Study Chair — Duke University Medical Center: Division of Rheumatology and Immunology
Locations (5):
- United States (5):
  - University of California San Francisco School of Medicine: Lupus Clinic and Rheumatology Clinical Research Center, San Francisco, California
  - University of Colorado School of Medicine: Division of Rheumatology, Aurora, Colorado
  - Brigham & Women's Hospital: Department of Medicine, Rheumatology, Immunology, Boston, Massachusetts
  - University of Michigan Health System: Department of Internal Medicine, Division of Rheumatology, Ann Arbor, Michigan
  - Duke University Medical Center: Division of Rheumatology and Immunology, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial
Access Criteria: Open access.
URL: http://www.immport.org/home

REFERENCES:
- See also: Immune Tolerance Network (ITN) — https://www.immunetolerance.org/
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait